CLINICAL TRIAL: NCT06261164
Title: Development and Use of a Population Pharmacokinetic Model of Amikacin and Vancomycin for the Optimization of Dosing Regimens in Critically Ill Patients on Different Modalities of Extracorporeal Hemoadsorption
Brief Title: Population Pharmacokinetic Model of Amikacin and Vancomycin in Critically Ill Patients
Status: Recruiting | Type: Observational
Sponsor: University Clinical Centre of Republic of Srpska (Other)
Responsible Party: Principal Investigator, Nikolina Spiric, MPharm, University Clinical Centre of Republic of Srpska
Other Study IDs: 01-19-373- 2/23
Record Dates: First submitted 2024-01-30; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients on hemodiafiltration with Cytosorb®
  Interventions: Device: Cytosorb® and Oxiris® adsorbents
- Patients on hemodiafiltration with Oxiris®
  Interventions: Device: Cytosorb® and Oxiris® adsorbents

INTERVENTIONS:
Device: Cytosorb® and Oxiris® adsorbents — The pharmacokinetic profile and the investigation of factors of pharmacokinetic variability of amikacin and vacnomycin in critically ill patients with a diagnosis of sepsis-like condition (SIRS), hospital-acquired sepsis and/or septic shock and who are on extracorporeal therapy with Cytosorb® and Oxiris® adsorbents.
  Other Names: Drugs' concentrations measurements

SUMMARY:
The object of the scientific research is the characterization of the pharmacokinetic profile and the investigation of factors of pharmacokinetic variability of amikacin and vacnomycin in critically ill patients with a diagnosis of sepsis-like condition (SIRS), hospital-acquired sepsis and/or septic shock and who are on extracorporeal therapy with Cytosorb® and Oxiris® adsorbents.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of SIRS, sepsis and/or septic shock,
* older than 18 years, who are being treated with amikacin and/or vancomycin,
* length of use of adsorbent at least 12 hours.

Exclusion Criteria:

* contraindication for hemodiafiltration with adsorbents,
* patients under the age of 18,
* terminal cancer patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult critically ill patients with a diagnosis of SIRS, sepsis and/or septic shock who are hospitalized in the Department of Medical Intensive Care Medicine
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Development of population pharmacokinetic model | One year
  Measurement of amikacin and vancomycine serum concentrations in several time points in order to gain pharmacokinetic profiles of previously mentioned drugs and to develop population pharmacokinetic model of amikacin and vancomycin by nonlinear modeling of combined effects in critically ill patients on veno-venous hemodiafiltration with two types of adsorbents.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolina Spiric, MPharm, Principal Investigator — University Clinical Centre of Republic of Srpska
Locations (1):
- Department of Medical Intensive Care Medicine, Banja Luka, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: No